CLINICAL TRIAL: NCT02181218
Title: A Multicenter Phase I Dose-finding and Preliminary Efficacy Study of the Histone Deacetylase Inhibitor Romidepsin (Istodax) in Combination With Gemcitabine (Gemzar), Oxaliplatin (Eloxatin), and Dexamethasone for the Treatment of Adults With Relapsed/Refractory Aggressive Lymphomas
Brief Title: Phase I Study of Romidepsin, Gemcitabine, Oxaliplatin, and Dexamethasone in Patients With Relapsed/Refractory Aggressive Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201407160
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse | interventions — romidepsin; Gemcitabine; Oxaliplatin; Dexamethasone; Calcium Dobesilate; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 0 (starting dose) (8 mg/m2 romidepsin) (Experimental): * Romidepsin will be administered intravenously (IV) over 2 hours on Days 2 and 8;
  * Gemcitabine IV over 30 minutes on Day 1
  * Oxaliplatin IV over 2 hours on Day 1
  * Dexamethasone orally on Days 1-4
  * Pegfilgrastim subcutaneously on Day 3
  * Drugs may be administered in any order on Day 1.
  * Each cycle is 21 days.
  * May continue on therapy for up to 8 cycles total if achieving adequate disease control (CR, PR, or stable disease) and without significant toxicity
  Interventions: Drug: Romidepsin; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Dexamethasone; Drug: Pegfilgrastim
- Dose Level 1 (10 mg/m2 romidepsin) (Experimental): * Romidepsin will be administered intravenously (IV) over 2 hours on Days 2 and 8;
  * Gemcitabine IV over 30 minutes on Day 1
  * Oxaliplatin IV over 2 hours on Day 1
  * Dexamethasone orally on Days 1-4
  * Pegfilgrastim subcutaneously on Day 3
  * Drugs may be administered in any order on Day 1.
  * Each cycle is 21 days.
  * May continue on therapy for up to 8 cycles total if achieving adequate disease control (CR, PR, or stable disease) and without significant toxicity
  Interventions: Drug: Romidepsin; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Dexamethasone; Drug: Pegfilgrastim
- Dose Level 2 (12 mg/m2 romidepsin) (Experimental): * Romidepsin will be administered intravenously (IV) over 2 hours on Days 2 and 8;
  * Gemcitabine IV over 30 minutes on Day 1
  * Oxaliplatin IV over 2 hours on Day 1
  * Dexamethasone orally on Days 1-4
  * Pegfilgrastim subcutaneously on Day 3
  * Drugs may be administered in any order on Day 1.
  * Each cycle is 21 days.
  * May continue on therapy for up to 8 cycles total if achieving adequate disease control (CR, PR, or stable disease) and without significant toxicity
  Interventions: Drug: Romidepsin; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Dexamethasone; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Romidepsin
  Other Names: Istodax®
Drug: Gemcitabine
  Other Names: GEMZAR®
Drug: Oxaliplatin
  Other Names: Eloxatin TM
Drug: Dexamethasone
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak® Taperpak®
Drug: Pegfilgrastim
  Other Names: Neulasta®

SUMMARY:
The purpose of this research study is to find the maximum tolerated dose of a drug called romidepsin when given with a treatment regimen called GemOxD. GemOxD is a routine treatment for certain types of lymphoma, and involves the administration of three drugs: gemcitabine, oxaliplatin, and dexamethasone. In addition to finding the maximum tolerated dose of romidepsin, the investigators want to look at the side effects of these drugs when given together, as well as how the lymphoma responds to this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign an informed consent form
* Age ≥ 18 at time of informed consent
* Diagnosis of one of the following:

  * relapsed/refractory peripheral T-cell lymphoma of any subtype including mycosis fungoides and Sézary syndrome of advanced stage (IIB-IVB)

    **for the expansion cohort:patients must have biopsy-proven T-cell lymphoma and measurable disease.
  * relapsed/refractory DLBCL (up to 6 DLBCL patients are allowed in the dose-escalation portion of the study)
  * relapsed/refractory HL

Note: extracorporeal photopheresis is NOT considered a systemic therapy for this study.

* Transplant eligible (as determined by referring physician) patients who have failed one prior salvage therapy or transplant ineligible (as determined by referring physician) patients who have failed one prior therapy
* ECOG performance status of ≤ 2
* Laboratory test results within the following ranges:

  * Absolute neutrophil count ≥ 1500/mm³
  * Platelet count ≥ 100,000/mm³
  * Total bilirubin ≤ 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
  * Creatinine < 2 mg/dL
  * Potassium ≥ 3.3 mmol/L or at/above the lower limit of normal for the performing laboratory
  * Magnesium ≥ 1.4 mg/dL or at/above the lower limit of normal for the performing laboratory.
* Negative serum pregnancy test for women of childbearing potential
* Washout time of at least 4 weeks for prior biological, chemotherapeutic, or radiotherapy

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would - in the opinion of the investigator - prevent the subject from signing the informed consent form
* Pregnant or lactating women
* Any medical condition or laboratory abnormalities, which - in the opinion of the investigator - places the subject at unacceptable risk, or confounds the ability to interpret data if he/she were to participate in the study
* Positive CSF cytology during staging, symptomatic leptomeningeal involvement, or parenchymal involvement of brain or spinal cord
* Prior allogeneic hematopoietic cell transplant
* Prior solid organ transplant
* Cirrhotic liver disease from any cause
* Known HIV infection
* Impaired cardiac function or clinically significant cardiac disease including any of the following:

  * Congenital long QT syndrome
  * Screening ECG with QTc interval ≥ 500 milliseconds
  * Myocardial infarction (MI) or unstable angina ≤ 6 months of C1D1; however, subjects with a history of MI between 6 and 12 months who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event would be eligible
  * Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV. In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
  * An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
  * Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (defined here as ventricular rate < 50 bpm); right bundle-branch block + left anterior hemi-block (bifasicular block)
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix 9) and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI History or presence of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), torsade de pointes, or cardiac arrest
  * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes
  * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria
  * Any cardiac arrhythmia requiring an anti-arrhythmic medication, excluding stable (i.e., at least 30 days from screening) doses of beta-blockers
* Concomitant use of drugs that may cause significant QT prolongation and/or torsades de pointes that cannot be discontinued or switched to a different medication prior to treatment
* Concomitant use of CYP3A4 inhibitors or inducers unless able to stop medication(s) prior to starting study treatment
* Patients who are unwilling to stop the use of herbal remedies while receiving study treatment
* Unable to accept blood product transfusions
* Men whose sexual partners are women of childbearing potential not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
* Concurrent malignancy requiring active therapy *Patients with localized prostate cancer having undergone surgery or radiation (field confined to ≤ 30% of marrow-bearing bone) at least 30 days prior to study treatment are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (recommended Phase II dose) | 37 months (completion of first cycle of all participants in study)
  Three participants will be treated at each dose level. If 0/3 patients experience dose limiting toxicity (DLT), 3 patients will be treated at the next dose level. If a DLT attributable to the treatment is experienced in 1 of 3 patients, three more patients (for a total of six participants) will be treated at that dose level. If no additional DLTs are observed at the expanded dose level (i.e. 1 of 6 with DLT), the dose will be escalated. Escalation will terminate as soon as two or more participants experience any DLT attributable to study combination, at a given dose level. If 2 or more DLTs occur at the starting dose level, a decreased dose level will be explored at dose level -1.
  There will be no more than 2 patients dosed for the first time within the same week, and patients in the next higher cohorts will not be enrolled until the last patient of the lower cohort has completed the DLT monitoring period, defined as 21 days after first dose of Cycle 1 therapy.

SECONDARY OUTCOMES:
Complete response rate | Up to 1 year from time of maximal response
  For study participants with relapsed/refractory peripheral T-cell lymphoma (PTCL), diffuse large b-cell lymphoma (DLBCL), and Hodgkin's lymphoma response will be assessed in accordance with the updated International Working Group (IWG) recommendations.
  For study participants with cutaneous t-cell lymphoma (CTCL), the Global Response Score established by the ISCL/USCLC/EORTC consensus panel will be used to assess response to treatment.
Partial response rate | Up to 1 year from time of maximal response
  For study participants with relapsed/refractory peripheral T-cell lymphoma (PTCL), diffuse large b-cell lymphoma (DLBCL), and Hodgkin's lymphoma response will be assessed in accordance with the updated International Working Group (IWG) recommendations.
  For study participants with cutaneous t-cell lymphoma (CTCL), the Global Response Score established by the ISCL/USCLC/EORTC consensus panel will be used to assess response to treatment.
Overall response rate | Up to 1 year from time of maximal response
  For study participants with relapsed/refractory peripheral T-cell lymphoma (PTCL), diffuse large b-cell lymphoma (DLBCL), and Hodgkin's lymphoma response will be assessed in accordance with the updated International Working Group (IWG) recommendations.
  For study participants with cutaneous t-cell lymphoma (CTCL), the Global Response Score established by the ISCL/USCLC/EORTC consensus panel will be used to assess response to treatment.
  Overall response rate = complete response + partial response
Progression free survival | Up to 1 year from time of maximal response
  Progression-free survival (PFS) will be defined as the time from registration until disease progression.
Duration of response | Up to 1 year from time of maximal response

CONTACTS AND LOCATIONS:
Overall Officials: Neha Mehta-Shah, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foley N, Riedell PA, Bartlett NL, Cashen AF, Kahl BS, Fehniger TA, Fischer A, Moreno C, Liu J, Carson KR, Mehta-Shah N. A Phase I Study of Romidepsin in Combination With Gemcitabine, Oxaliplatin, and Dexamethasone in Patients With Relapsed or Refractory Aggressive Lymphomas Enriched for T-Cell Lymphomas. Clin Lymphoma Myeloma Leuk. 2025 May;25(5):328-336. doi: 10.1016/j.clml.2024.11.015. Epub 2024 Dec 4. PMID 39725584
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu